CLINICAL TRIAL: NCT05321550
Title: De Nociceptieve Flexie Reflex Als Diagnostische Test Voor Centrale Sensitisatie
Brief Title: The Nociceptive Flexion Reflex as a Diagnostic Tool of Central Sensitization
Acronym: NFR-CS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-5159
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Central Sensitisation; Fibromyalgia; Neck Pain; Low Back Pain; Whiplash
MeSH Terms: conditions — Fibromyalgia; Neck Pain; Low Back Pain; Whiplash Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Fibromyalgia patients: Fibromyalgia patients diagnosed according to the 2010 ACR-criteria
- Neck pain patients: * Patients with non-specific, idiopathic neck pain complaints
  * Patients with neck pain complaints of traumatic origin type whiplash grade 1 (pain, stiffness or tenderness of the neck and no objective physical abnormalities) and grade 2 (neck complaints and musculoskeletal disorders such as reduced range of motion and tender pain points) according to the Quebec Task Force on Whiplash Associated Disorders
- Low back pain patients: Patients with non-specific, idiopathic back pain complaints
- Healthy controls: Age, sex and BMI-matched healthy controls

SUMMARY:
This experimental study will investigate whether the decreased NFR threshold and increased NFR temporal summation, which are frequently observed in chronic pain patients, are only symptomatic manifestations that occur in the involved limb and indicate peripheral sensitization or generalized manifestations that are also present in the non-involved limbs and thus indicate central sensitization. To gain an idea of the presence of central sensitization, this study will also investigate whether there are increased perception and decreased pain thresholds in response to electrical, thermal, and mechanical stimulation, as well as whether there is a decreased conditioned pain modulation. To investigate this, it is essential to examine different pain populations and locations, in particular, acute pain versus chronic pain populations to compare peripheral versus central sensitization, respectively. Recently, our research group has shown that patients with a traumatic origin of chronic neck pain (chronic whiplash-associated disorders) show central sensitization in contrast to patients with a non-traumatic origin (chronic idiopathic neck pain) who demonstrate only indications for peripheral sensitization. Therefore, this study will also distinguish between complaints of traumatic and non-traumatic origin.

The measurements will be performed at different locations, namely the lower and upper limbs. To determine whether the differences depend on the measurement location (= location where experimental nociceptive stimulation is administered) and symptom location (= location of clinical nociceptive stimulation), different patient populations will be compared with each other, as well as with a healthy control population. In acute and chronic whiplash patients and patients with acute and chronic idiopathic neck pain complaints, the complaints are primarily localized in the upper limb. It is hypothesized that in chronic neck pain patients (both whiplash and idiopathic neck pain patients) abnormal values are found in both the upper and lower limbs compared to the healthy controls due to central sensitization. In acute neck pain patients (both whiplash and idiopathic neck pain) only abnormal values in the arm are expected and not in the leg as a result of peripheral sensitization. It is hypothesized that patients with neck pain of traumatic origin will show a stronger sensitization than those with neck pain of non-traumatic origin. In acute and chronic low back pain patients, the complaints are primarily localized in the lower body quadrant. As a result of central sensitization in the chronic low back pain patients, abnormal values are expected in both the upper and lower limbs, while only abnormal values in the leg are expected as a result of peripheral sensitization in the acute low back pain patients. Finally, this study will investigate whether chronic low back and neck pain patients show a similar pattern of central sensitization as fibromyalgia patients, a population with generalized complaints that are primarily attributed to central sensitization.

ELIGIBILITY:
Inclusion Criteria Fibromyalgia patients:

- diagnosed according to 2010 ACR-criteria

Inclusion Criteria neck pain patients:

- having idiopathic neck pain complaints or having grade 1 (pain, stiffness or tenderness of the neck and without objective physical abnormalities) or grade 2 (neck complaints and musculoskeletal disorders such as decreased range of motion and tender pain points) according to the Quebec Task Force on Whiplash Associated Disorders

Inclusion Criteria low back pain patients:

- having idiopathic low back pain complaints

Inclusion Criteria healthy controls:

* no history of serious pain complaints (e.g. severe migraine, fibromyalgia, etc.)
* no low back or neck pain complaints with an intensity of ≥2/10 on a visual analogue scale in the past year and of such severity that the daily activities were disrupted and a (para)medic was consulted

Exclusion Criteria:

* history of severe respiratory (e.g. cystic fibrosis), orthopedic (e.g. whiplash trauma), neurological (e.g. cerebrovascular incident), cardiovascular (e.g. severe hypertension), or endocrinological (e.g. diabetes) disorders
* recent psychological trauma (e.g. post-traumatic stress disorder)
* history of spinal surgery (e.g. lumbar discectomy), spinal trauma (e.g. vertebral fracture), or severe spinal deformities (e.g. spondylolisthesis)
* BMI ≥35 (due to potential difficulties in obtaining an NFR in severely overweight individuals)
* having pacemakers and defibrillators (absolute exclusion criteria for electrical stimulus stimulation, i.e. TENS)
* pregnancy, lactation, or within 1 year postpartum

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Fibromyalgia patients (n=30) diagnosed according to the 2010 ACR-criteria
  * Patients with non-specific, idiopathic neck pain complaints which are acute (n=30) or chronic (n=30)
  * Patients with neck pain complaints of traumatic origin type whiplash grade 1 (pain, stiffness or tenderness of the neck and no objective physical abnormalities) and grade 2 (neck complaints and musculoskeletal disorders such as reduced range of motion and tender pain points) according to the Quebec Task Force on Whiplash Associated Disorders which is acute (n=30) or chronic (n=30)
  * Patients with non-specific, idiopathic back pain complaints which are acute (n=30) or chronic (n=30)
  * Healthy controls (n=30) matched based on age, sex and BMI
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Quantitative sensory testing (QST) - electrical detection threshold | Baseline
  Determination of sensory detection thresholds in response to electrical stimuli which are delivered transcutaneously over the n. suralis and n. medianus, recorded in mA.
Quantitative sensory testing (QST) - electrical pain threshold | Baseline
  Determination of sensory pain threshold in response to electrical stimuli which are delivered transcutaneously over the n. suralis and n. medianus, recorded in mA.
Quantitative sensory testing (QST) - thermal detection threshold | Baseline
  Determination of sensory detection thresholds in response to thermal stimuli which are delivered to the skin using a thermode, recorded in °C:
  * cold detection threshold
  * warmth detection threshold
Quantitative sensory testing (QST) - thermal pain threshold | Baseline
  Determination of sensory pain thresholds in response to thermal stimuli which are delivered to the skin using a thermode, recorded in °C:
  * cold pain threshold
  * heat pain threshold
Quantitative sensory testing (QST) - discrimination between thermal stimuli | Baseline
  Determination of the number of paradoxical heat sensations in response to alternating cold and warm stimuli delivered to the skin using a thermode.
Quantitative sensory testing (QST) - tactile detection threshold | Baseline
  Determination of tactile detection threshold, assessed using Von Frey monofilaments, recorded in mN
Quantitative sensory testing (QST) - mechanical pain threshold | Baseline
  Determination of mechanical pain threshold, assessed using pinprick stimulators, recorded in mN
Quantitative sensory testing (QST) - sensitivity to pressure stimuli | Baseline
  Determination of pressure pain threshold, assessed using pressure algometry, recorded in kg
Quantitative sensory testing (QST) - temporal summation of electrical stimuli | Baseline
  Determination of temporal summation in response to electrical stimuli delivered transcutaneously over the skin of the n. suralis and n. medianus.
  The numerical pain rating in response to these stimuli (range 0 - 100) will be recorded.
Quantitative sensory testing (QST) - spinal hyperexcitability | Baseline
  Determination of spinal hyperexcitability using the nociceptive flexion reflex (NFR; sensitization of spinal cord neurons), recorded in mA
Quantitative sensory testing (QST) - temporal summation of spinal hyperexcitability | Baseline
  Determination of temporal summation of the nociceptive flexion reflex (NFR; sensitization of spinal cord neurons), recorded using a numeric pain rating scale (range 0 - 100)
Quantitative sensory testing - conditioned pain modulation | Baseline
  Determination of condition pain modulation (aka. pain inhibits pain) by means of a heterotopic noxious counterstimulation paradigm. Test stimuli comprise of pressure pain threshold assessments and application of a heat stimulus (using a thermode) corresponding to a temperature eliciting a visual analog scale rating of 5/10. Test stimuli will be applied before, during and after the conditioning stimulus which is the immersion of the hand in a hot circulating water bath of 45.5°C.

SECONDARY OUTCOMES:
Central sensitization inventory | Baseline
  Self-report measure of signs and symptoms associated with central sensitization
Douleur Neuropathique 4 Questionnaire | Baseline
  Clinician administered questionnaire for evaluation of signs and symptoms associated with neuropathic pain
Pain catastrophizing scale | Baseline
  Self-report measure of pain perceptions and cognitions
Pain vigilance and awareness questionnaire | Baseline
  Self-report measure assessing preoccupation with and attention to pain
Tampa scale for kinesiophobia | Baseline
  Self-report measure assessing fear of movement
International physical activity questionnaire | Baseline
  Self-report measure of physical activity in preceeding 7 days
Patient-reported outcomes measurement information system - physical functioning | Baseline
  Self-report measure of health-related domains relating to physical functioning
Patient-reported outcomes measurement information system - anxiety | Baseline
  Self-report measure of health-related domains relating to anxiety
Patient-reported outcomes measurement information system - depression | Baseline
  Self-report measure of health-related domains relating to depression
Patient-reported outcomes measurement information system - fatigue | Baseline
  Self-report measure of health-related domains relating to fatigue and sleep disruption
Patient-reported outcomes measurement information system - participation | Baseline
  Self-report measure of health-related domains relating to participation in social activities
Patient-reported outcomes measurement information system - pain interference | Baseline
  Self-report measure of health-related domains relating to pain interference
Injustice Experience Questionnaire | Baseline
  Self-report measure of perceived injustice
Pain Disability Index | Baseline
  Self-report measure of pain-related disability

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Van Oosterwijck, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided